CLINICAL TRIAL: NCT05831033
Title: Safety and Efficacy of an Autologous Tumor Infiltrating Lymphocyte (TIL) Therapy in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiaotong University School of Medicine (Unknown); RenJi Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Director of Medical Oncology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101T1
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: Cell Therapy; Autologous Adoptive Cell Therapy; Tumor Infiltrating Lymphocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BEN101 (Experimental): BEN101 infusion single dose level between 1x10^9 to 1x 10^11，not lower than 1×10^9 cells, final dose is affected by the starting amount of TILs cells isolated from the tumor tissue sample.
  Interventions: Biological: BEN101

INTERVENTIONS:
Biological: BEN101 — Lymphodepletion regimen：Cyclophosphamide 250mg/ m2/day x 3 days (day -4, -3，-2) , Fludarabine 25mg/ m2/day x 2 days (day-4, -3) , Paclitaxel 100mg/ m2/day -3. The lymphodepletion regimen could be adjusted by the treating physician according to patient's disease condition.
  BEN101 infusion： Single dose level between 1x10^9 to 1x 10^11，not lower than 1×10^9 cells, final dose is affected by the starting amount of TILs cells isolated from the tumor tissue sample.
  IL-2：Administer 8-16 hr after TIL infusion. 600,000 IU/kg intravenously over 15-20 mins every 12 hours. It is recommended to start with high dose; and de-escalate based on tolerability, up to 5 days. IL-2 administration will be terminated if unacceptable toxicities occur.

SUMMARY:
Multicenter, single arm, non-randomized, prospective, open label, interventional study evaluating adoptive cell therapy (ACT) with autologous tumor infiltrating lymphocytes (TIL) infusion (BEN101) followed by IL-2 after a non-myeloablative (NMA) lymphodepletion preparative regimen for the treatment of patients with recurrent and/or metastatic solid tumor.

DETAILED DESCRIPTION:
BEN101 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, for the treatment of patients with recurrent and/or metastatic solid tumor. The cell transfer therapy used in this study involves patients receiving a NMA lymphocyte depleting preparative regimen, followed by infusion of autologous TIL followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion criteria

1. Be able and willing to provide written informed consent, and to comply with all requirements of study participation (including all study procedures).
2. Age: 18 - 75 years.
3. Histological or cytological diagnosis of advanced metastatic solid tumors.
4. Progression on standard therapy, or intolerance to, refusal or unable to benefit from standard therapy according to investigator's judgement.
5. At least one resectable lesion (or aggregate of lesions) of a minimum 15 mm in diameter post-resection; or core biopsy (aggregate of around 1 gram or two 18G puncture needles).
6. At least one measurable target lesion, as defined by RECIST v1.1.Lesions in previously irradiated areas (or other local therapy) should not be selected as target lesions, unless treatment was ≥ 3 months prior to screening, and there has been demonstrated disease progression in that particular lesion.
7. ECOG performance status of 0 or 1.
8. Life expectancy of at least 3 months.
9. Adequate organ and marrow function (hematology, renal, hepatic and coagulation).

   1. Absolute neutrophil count (ANC) ≥ 1.0×10^9/L.
   2. Hemoglobin (Hb) ≥ 80 g/L.
   3. Platelet ≥ 75×10^9/L.
   4. Sufficient coagulation: APPT<40 and INR<1,5.
   5. Creatinine clearance (CrCL) ≥45 mL/min or serum creatinine ≤1.5mg/dL was estimated using the Cockcroft-Gault formula.
   6. Serum alanine transaminase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) and aspartate transaminase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤ 3 times the upper limit of normal (ULN); patients with liver metastasis ≤ 5 times ULN.
   7. Estimated creatinine clearance (eCrCl) ≥ 40 mL/min using the Cockcroft-Gault formula.
   8. Total bilirubin ≤ 1.5 times ULN.
   9. Patients with Gilbert's syndrome must have a total bilirubin ≤ 1.5 times ULN.
   10. Patients with left ventricular ejection fraction (LVEF) ≥50% or New York Heart Association (NYHA) functional classification ≤ Class 1.
   11. Patients with pulmonary function test (forced expiratory volume in 1 second FEV1) ≥75%.

Exclusion criteria

1. Patients who have received an organ allograft or prior cell transfer therapy.
2. Patients who have a history of hypersensitivity to any component or excipient of study drugs.
3. Patients who have active central nervous system (CNS) metastases（except stable brain metastases without hormone dependence or drug treatment within 3 months before enrollment）.
4. Patients who have active medical illness(es) that would pose increased risk for study participation, including: active systemic infections requiring systemic antibiotic therapy, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune system.
5. Active hepatitis C subjects (Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive), human immunodeficiency virus (HIV) antibody positive; syphilis primary screening antibody positive; untreated active hepatitis B subjects (hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA quantitative test greater than ULN), hepatitis B subjects need to receive anti-HBV treatment during the study period.
6. Previous history of immunodeficiency (any form, primary or acquired), current long-term use of systemic corticosteroids or other immunosuppressants. Patients receiving steroids as replacement therapy for adrenocortical insufficiency at ≤ 10 mg/day of prednisone or other steroid equivalent may be eligible.
7. Patients who have had another primary malignancy within the previous 3 years (with the exception of carcinoma in situ of the breast, cervix, or bladder; localized prostate cancer; and non-melanoma skin cancer that has been adequately treated).
8. Patients who have received a live or attenuated vaccine within 28 days before signing the informed consent.
9. Received other cell therapy products in the past.
10. History of Grade ≥3 immune mediated AE (including AST/ALT elevations that where considered drug related and cytokine release syndrome) that was considered related to prior immune modulatory therapy (eg, immune checkpoint inhibitors, co-stimulatory agents, etc.) and required immunosuppressive therapy.
11. Patients who are pregnant or breastfeeding.
12. Before enrollment, adverse event due to any previous treatment or surgery which had not recovered to ≤ Grade 1 (according to CTCAE V5.0); except: alopecia, peripheral neuropathy ≤ grade 2, events that remain stable during supportive therapy (such as stable hypothyroidism with hormone replacement therapy), or other events that have no safety risk as assessed by the investigator.
13. Patients who do not consent to the use of medically approved contraceptive methods during the study.
14. Patients whose cancer requires immediate attention or who in the investigator's judgement is not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 6 month
  Adverse events according to CTCAE v5.0, Treatment Emergent Adverse event (TEAE) >=grade 3; Treatment related adverse event (TRAE).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Proportion of patients with response to evaluate efficacy parameters such as Objective Response Rate (ORR) using RECIST v1.1 as assessed by the Investigator
Disease Control Rate (DCR） | Up to 24 months
  Proportion of patients with response per response to evaluate efficacy parameters such as Disease Control Rate (DCR) using RECIST v1.1 as assessed by the Investigator
Duration of response (DOR) | Up to 24 months
  To evaluate efficacy parameters such as Duration of Response (DOR) using RECIST v1.1 as assessed by the Investigator
Progression free survival (PFS) | Up to 24 months
  The time length between BEN101 infusion and confirmed subsequent disease progression according to RECIST 1.1
Overall survival (OS) | Up to 24 months
  The length of time from the date of the start of BEN101 treatment that the patients are still alive

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Doctor, Principal Investigator — Shanghai General Hospital, Fudan University Shanghai Cancer Center; Wen Di, Doctor, Principal Investigator — RenJi Hospital; Wei Xue, Doctor, Principal Investigator — RenJi Hospital; Weiyi Huang, Master, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No
to publish papers